CLINICAL TRIAL: NCT00156767
Title: Adrenal Function in Critical Illness
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050013; 05-CH-0013
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-03-28

CONDITIONS: Adrenal Insufficiency
Keywords: ACTH; Cortisol; Natural History
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Bone Marrow Transplant: Patients enrolled in an NCI protocols for bone marrow transplant for breast cancer using prednisone treatment.
- Cirrhosis: Adults on NIDDK protocol 91-DK-0213 with evidence of chronic liver disease with class A or B cirrhosis secondary to viral hepatitis
- Critical Care: Patients with a diagnosis of sepsis by the primary clinical provider in the Emergency room of ICU
- Healthy Volunteer: Healthy adult volunteers
- Known Adrenal Insufficiency: patients with known diagnosis of Adrenal Insufficiency
- Nephrotic Syndrome: Adults enrolled in NIDDK protocols with diagnosis of nephrotic syndrome
- Post Surgical Treatment for Cushings: Patients with transient adrenal insufficiency secondary to successful surgical treatment of cushing's syndrome

SUMMARY:
An appropriate hypothalamic-pituitary-adrenal (HPA) axis response is required to survive critical illness. Primary adrenal insufficiency, relative adrenal insufficiency, tissue resistance to glucocorticoids, ACTH deficiency and immune-mediated inhibition of the HPA axis may impair the secretion or action of glucocorticoids in critically ill patients. Adrenal insufficiency is estimated to occur in up to 77% of critically ill patients, but currently, there is no consensus on the diagnostic criteria for adrenal insufficiency in this setting, and standard testing does not discriminate among the aforementioned factors. We will study the incidence and natural history of adrenal insufficiency in critically ill patients to further define adrenal insufficiency and provide data to develop diagnostic tests. Clinical features and outcomes will be correlated with laboratory measurements of hormones, cytokines and glucocorticoid action. Healthy volunteers will undergo cortrosyn tests with measurement of free cortisol levels to develop a normative range for this endpoint.

<TAB>

Previous glucocorticoid use, if prolonged and supraphysiologic, also inhibits the HPA and can result in adrenal insufficiency. Patients with short intermittent courses of glucocorticoid administration have not been studied well, and may also be at risk. To gain further information about this group, patients receiving pulse glucocorticoid doses as part of bone marrow transplant regimens at the Clinical Center will also be studied.

DETAILED DESCRIPTION:
An appropriate hypothalamic-pituitary-adrenal (HPA) axis response is required to survive critical illness. Primary adrenal insufficiency, relative adrenal insufficiency, tissue resistance to glucocorticoids, ACTH deficiency and immune-mediated inhibition of the HPA axis may impair the secretion or action of glucocorticoids in critically ill patients. Adrenal insufficiency is estimated to occur in up to 77 percent of critically ill patients, but currently, there is no consensus on the diagnostic criteria for adrenal insufficiency in this setting, and standard testing does not discriminate among the aforementioned factors. We will study the incidence and natural history of adrenal insufficiency in critically ill patients to further define adrenal insufficiency and provide data to develop diagnostic tests. Clinical features and outcomes will be correlated with laboratory measurements of hormones, cytokines and glucocorticoid action. Healthy volunteers will undergo cortrosyn tests with measurement of free cortisol levels to develop a normative range for this endpoint. Patients with known adrenal insufficiency will also be studied to help determine the clinical utility of diagnostic tests among these different groups. Previous glucocorticoid use, if prolonged and supraphysiologic, also inhibits the HPA axis and can result in adrenal insufficiency. Patients with short intermittent courses of glucocorticoid administration have not been studied well, and may also be at risk. To gain further information about this group, patients receiving pulse glucocorticoid doses as part of bone marrow transplant regimens at the Clinical Center will also be studied.

ELIGIBILITY:
* CRITERIA FOR ALL ARMS OF STUDY:

Women of reproductive age will also undergo a pregnancy test (urine hCG) prior to starting the testing procedure. If the woman is determined to be pregnant, she will not be able to participate in this study.

CRITICAL CARE COMPONENT:

INCLUSION CRITERIA:

Diagnosis of sepsis by the primary clinical provider in the ICU.

Diagnosis of the above is based on diagnostic criteria for sepsis as defined by the 2001 SCCM/ESICM/ACCP/ATS/SIS International Sepsis Definitions Conference as listed below:

Infection, documented or suspected, and some of the following:

General variables

* Fever (core temperature greater than 38.3 C)
* Hypothermia (core temperature greater than 36C)
* Heart Rate greater than 90 min or greater than 2 SD above the normal value for age
* Tachypnea
* Altered mental status
* Significant edema or positive fluid balance (greater than 20ml/kg over 24 hours)
* Hyperglycemia (plasma glucose greater than 120 mg/dl) in the absence of diabetes

Inflammatory variables

* Leukocytosis (WBC count greater than 12,000 uL)
* Leukopenia (WBC count less than 4000 uL)
* Normal WBC count with greater than 10 percent immature forms
* Plasma C-reactive protein greater than 2 SD above the normal value
* Plasma procalcitonin greater than 2 SD above the normal value

Hemodynamic variables

* Arterial hypotension (SBP less than 90mm Hg, MAP less than 70, or an SBP decrease greater than 40 mm Hg in adults or less than 2 SD below normal for age)
* SvO2 greater than 70 percent
* Cardiac Index greater than 3.5L min(-1) M(-23)

EXCLUSION CRITERIA:

Pregnancy

Age less than 15 years at the Clinical Center; age less than 18 years at Georgetown or Suburban Hospitals

On glucocorticoids or megace within two weeks of admission unless using more than one of the following medications, patients taking inhaled corticosteriods (less than 1.5 mg/day budesonide, beclomethasone dipropionate and triamcinolone acetonide and less thab 0.75 mg/day for fluticasone propionate) or intranasal corticosteriods will not be excluded.

Patients who have received chronic steroid suppressive medications, i.e. etomidate, ketoconazole (Patients receiving etomidate for intubation purposes as a one time dose will not be excluded)

End stage renal or liver disease (creatinine clearance estimated as less than 20 cc/min by the cockcroft-gault equation: (140 - age) times lean body weight (kg)/ pCr (mg/dl) times 72, in patients with stable renal function; patients requiring dialysis; acute or fulminant hepatitis, alcoholic hepatitis, chronic severe hepatitis, severe obstructive hepatitis, severe coagulopathy, extrahepatic manifestations of ESLD, i.e. hypoxia, cardiomyopathy, acute renal failure)

Known or anticipated blood withdrawal within 6 weeks that exceeds the NIH guidelines of 450 l/six weeks in adults or 7 ml/kg/six weeks in children.

BONE MARROW TRANSPLANT COMPONENT:

INCLUSION CRITERIA:

Participation in a Clinical Center bone marrow transplant protocol for breast cancer (generally Allogeneic Breast Protocol 2: Phase 1 Trial of T cell Exchange with Th2/Tc2 Cells for Allogeneic Stem Cell Transplantation after Reduced Intensity Conditioning for Metastatic Breast Cancer), or for hematologic malignancy (generally either: T-cell depleted, reduced intensity allogeneic stem cell transplant from haploidentical related donors for hematologic malignancies: A sequential dose escalation study of donor Th2/Tc2 cells or Th2, Sirolimus in Allogeneic HSCT.

Agreement from the oncologist PI that the patient may participate in this protocol.

EXCLUSION CRITERIA:

The presence of any contraindication to insulin tolerance testing-e.g.cardiovascular or cerebrovascular disease or any seizure history.

Pregnancy

Age less than 15 years

End stage renal or liver disease as defined under the critical care section

Known or anticipated blood withdrawal within 6 weeks that exceeds the NIH guidelines of 450 ml/six weeks in adults.

HEALTHY VOLUNTEER COMPONENT:(Closed to recruitment)

INCLUSION CRITERIA:

Adults aged at least 18 years will be recruited.

EXCLUSION CRITERIA:

Severe hepatic, renal, cardiac, psychiatric or neurological illnesses

More than two weeks of oral antifungal or glucocorticoid medications or near daily use of topical glucocorticoids with broken skin. Frequent use of topical antifungal agents will be considered on a case-by-case basis.

Pregnancy

KNOWN ADRENAL INSUFFICIENCY COMPONENT:

INCLUSION CRITERIA:

Documented longstanding primary or secondary adrenal insufficiency

EXCLUSION CRITERIA:

Pregnancy

TRANSIENT ADRENAL INSUFFICIENCY COMPONENT:

INCLUSION CRITERIA:

Recent uncomplicated successful transsphemoidal surgery for Cushing s disease with serum cortisol level less than 5 micro g/dl

TRANSIENT ADRENAL INSUFFICIENCY COMPONENT:

EXCLUSION CRITERIA:

Supra physiologic dosing of glucocorticoids as a treatment for another underlying medical disorder or surgical complication

Pregnancy

CIRRHOSIS AND NEPHROTIC SYNDROME COMPONENT:

Adults aged at least 18 years will be recruited.

CIRRHOSIS

INCLUSION CRITERIA:

* Participation in an active NIDDK protocol entitled: Evaluation of patients with liver disease (91-DK-0214), with evidence of chronic liver disease
* Agreement from the hepatologist PI that the patient may participate in this protocol.
* Child-Pugh class A or B cirrhosis secondary to viral hepatitis
* Absence of other significant medical illnesses that might interfere with prolonged follow-up evaluation
* Normal renal function (creatinine clearance estimated as > 60 ml/min by the Modified Diet in Renal Disease (MDRD) equation and reported through our Clinical Research Information System (CRIS)).

EXCLUSION CRITERIA:

* History of the use of glucocorticoid therapy or medications that are known to interfere with HPA axis function within the past 6 months
* Current symptoms of adrenal insufficiency (nausea, vomiting, weight loss, lightheadedness, unusual fatigue, salt craving, etc.).
* Evidence of moderate-severe medical illness attributable to obstructive sleep apnea, heart or pulmonary failure, or active malignancy will be excluded.
* Pregnancy
* Known or anticipated blood withdrawal within 6 weeks that exceeds the NIH guidelines of 450 ml/six weeks in adults.

NEPHROTIC SYNDROME:

INCLUSION CRITERIA:

* Participation in one of three active NIDDK protocols entitled: Rituximab plus cyclosporine in idiopathic membranous nephropathy (09-DK-0223), the Nephrotic Syndrome Study Network (Neptune) (11-DK-0023), or Pathogenesis of Glomerulosclerosis Study (94-DK-0127) with previously documented proteinuria >3.5g/day for 2 months or more or protein/creatinine ratio of 2.0 g/g on at least 2 occasions
* Agreement from the nephrologist PI that the patient may participate in this protocol. Estimated GFR greater than or equal to 30 ml/min based on the MDRD equation and reported through CRIS.
* Normal liver function as defined by normal liver function tests and no known history of liver disease.

EXCLUSION CRITERIA:

* History of the use of glucocorticoid therapy or medications that are known to interfere with HPA axis function within the past 6 months
* Current symptoms of adrenal insufficiency (nausea, vomiting, weight loss, lightheadedness, unusual fatigue, salt craving, etc.).
* Evidence of moderate-severe medical illness attributable to obstructive sleep apnea, heart or pulmonary failure, or active malignancy will be excluded.
* Pregnancy
* Known or anticipated blood withdrawal within 6 weeks that exceeds the NIH guidelines of 450 ml/six weeks in adults.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NIH patients with Cushing's syndrome, adrenal insufficiency, hepatitis, nephrotic syndrome surrounding community healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2004-11-12 (Actual)

PRIMARY OUTCOMES:
Cortisol | after ACTH
  cortisol increase

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Abraham SB, Abel BS, Sinaii N, Saverino E, Wade M, Nieman LK. Primary vs secondary adrenal insufficiency: ACTH-stimulated aldosterone diagnostic cut-off values by tandem mass spectrometry. Clin Endocrinol (Oxf). 2015 Sep;83(3):308-14. doi: 10.1111/cen.12726. Epub 2015 Mar 20. PMID 25620457
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-CH-0013.html